CLINICAL TRIAL: NCT01275391
Title: cSBIRT to Reduce Teen Tobacco, Alcohol and Drug Use
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This project was not funded.
Sponsor: Boston Children's Hospital (Other)
Collaborators: Pearl Network (Network)
Responsible Party: Principal Investigator, John R Knight, MD, Associate Professor of Pediatrics, Harvard Medical School; Senior Associate in Medicine; Associate in Psychiatry, Director, Center for Adolescent Substance Abuse Research, Boston Children's Hospital, Boston Children's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RFADEcSBIRT
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Tobacco Abuse; Alcohol Abuse; Drug Abuse
Keywords: Tobacco use; Alcohol abuse; Drug abuse; Substance use; Prevention; Brief intervention; Screening; Adolescents
MeSH Terms: conditions — Tobacco Use Disorder; Alcoholism; Substance-Related Disorders; Tobacco Use | interventions — Crisis Intervention; Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment as Usual Group 1 (No Intervention): Participants will receive treatment as usual and will complete a baseline and 1-month post-visit assessment
- Treatment as Usual Group 2 (No Intervention): Participants will receive treatment as usual and complete only the 1-month post-visit assessment
- Intervention Group 1 (Experimental): Computer Screening, Brief Intervention, Referral toTreatment. Participants will receive the intervention and complete a baseline and 1-month post-visit assessment
  Interventions: Behavioral: Computer Screening, Brief Intervention, Referral toTreatment
- Intervention Group 2 (Experimental): Computer Screening, Brief Intervention, Referral toTreatment Participants will receive the intervention and complete only the 1-month post-visit assessment
  Interventions: Behavioral: Computer Screening, Brief Intervention, Referral toTreatment

INTERVENTIONS:
Behavioral: Computer Screening, Brief Intervention, Referral toTreatment — A computerized screening for tobacco, alcohol and drug use accompanied by 10-15 pages of health information regarding the risks of tobacco, alcohol and drug use. This is followed by a brief conversation with the primary care provider regarding the health risks of tobacco, alcohol and drug use and a referral to treatment for those at high risk of substance use problems.
  Other Names: Brief Advice; SBIRT; Screen and Brief Advice
  Arms: Intervention Group 1; Intervention Group 2

SUMMARY:
In this project we will conduct a pilot study of a brief intervention to reduce teen tobacco, alcohol and drug use that primary care dental practitioners can provide in their offices.

DETAILED DESCRIPTION:
The goal of this project is to prepare for a large multi-site comparative effectiveness trial of a behavioral intervention, computer-facilitated Screening, Brief Intervention, and Referral to Treatment (cSBIRT) system that targets tobacco, alcohol, and drug use among adolescent dental patients. This enhanced computerized screening system includes: (1) screening, feedback, and provider talking points for tobacco and non-medical use of prescription drugs, (2) an interactive 2-part Motivational Enhancement Therapy module for adolescents at highest risk to complete from home, and (3) technological extenders (TEs), which are computer-generated messages that the provider sends to adolescents during the months following the clinic visit to reinforce the effect of the intervention over time.

ELIGIBILITY:
Inclusion Criteria:

* 12-21 years of age
* arriving for routine care to dental office

Exclusion Criteria:

* dentally, medically, or psychologically unstable at the time of the visit
* cannot read or understand English at a 6th grade level
* unavailable for 1-month post-visit assessment

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Percent days abstinent of tobacco, alcohol and drugs | Past 90 days

SECONDARY OUTCOMES:
Prevalence of tobacco, alcohol and drug use | Past 90 days

CONTACTS AND LOCATIONS:
Overall Officials: John R. Knight, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holliday R, Hong B, McColl E, Livingstone-Banks J, Preshaw PM. Interventions for tobacco cessation delivered by dental professionals. Cochrane Database Syst Rev. 2021 Feb 19;2(2):CD005084. doi: 10.1002/14651858.CD005084.pub4. PMID 33605440
- See also: web site of the Center for Adolescent Substance Abuse Research at Children's Hospital Boston — http://www.ceasar.org